

SPONSOR: ZMS

PROTOCOL: ZMS-1600-Blood Loss Detection

# CLINICAL PROTOCOL ZMS-1600-Blood Loss Detection NCT#05463198 16-NOV-2022




SPONSOR: ZMS


#### **CLINICAL PROTOCOL**

| TITLE | Evaluation of Physiological Zynex Fluid Monitoring Sys | Variables and Detection of Bl<br>stem, Model CM-1600 | ood Loss Using the |
|---|---|---|---|
| PROTOCOL | ZMS-1600-Blood Loss Dete | ection | |
| SPONSOR | Zynex Monitoring Solution<br>9555 Maroon Circle<br>Englewood, CO 80112 | s (ZMS) | |
| PROTOCOL VERSION | 2.0 | | |
| DOCUMENT REVIEW<br>& APPROVAL | | | |
| Sponsor Representative: | | | |
| | | Signature | Date |
| Sponsor Representative: | | | |
| | | Signature | Date |



SPONSOR: ZMS




SPONSOR: ZMS


| | PROTOCOL SIGNATURE PAGE |
|---|---|
| TITLE PROTOCOL SPONSOR | Evaluation of Physiological Variables and Detection of Blood Loss Using the Zynex Fluid Monitoring System, Model CM-1600 ZMS-1600-Blood Loss Detection Zynex Monitoring Solutions (ZMS) 9555 Maroon Circle Englewood, CO 80112 |
| PROTOCOL VERSION | 2.0 |
| Principal Investigator (PI): | |
| | PI Printed Name |
| • | PI Signature |
| - | Date (DD-MMM-YYYY) |



SPONSOR: ZMS


| PROTOCOL AMENDMENT HISTORY | | |
|---|---|---|
| Version<br>Number | Description of Change(s) | Reason for Change |
| 1.0 | Initial protocol; no changes | N/A |
| 2.0 | Section 9.1 and throughout: Increase in sample size to 500 subjects | Additional subjects required to support statistical analyses. |
| | [This space is intentionally | eleft blank] |



SPONSOR: ZMS


#### **TABLE OF CONTENTS**

| 1 | INT | RODUCTION | 10 |
|---|---|---|---|
| | 1.1 | CLINICAL RATIONALE | 11 |
| 2 | INV | ESTIGATIONAL PLAN | 11 |
| | 2.1 | OBJECTIVES | 11 |
| | 2.2 | STUDY DURATION | 11 |
| | 2.3 | STUDY DESIGN | 11 |
| | 2.4 | STUDY ENDPOINTS | 11 |
| 3 | STU | IDY DEVICES | 12 |
| | 3.1 | FLUID MONITORING SYSTEM, MODEL CM-1600 | 12 |
| | 3.1. | 1 DEVICE DESCRIPTION | 12 |
| | 3.1. | 2 DEVICE DESIGN AND COMPONENTS | 12 |
| | 3.1. | 3 PRINCIPLES OF OPERATION | 12 |
| | 3.1. | 4 INDICATIONS FOR USE | 12 |
| | 3.1. | 5 INTENDED USE | 12 |
| 4 | SUB | BJECT POPULATION AND SELECTION | 13 |
| | 4.1 | POPULATION AND ANTICIPATED NUMBER OF SUBJECTS | 13 |
| | 4.2 | SUBJECT INCLUSION CRITERIA | 13 |
| | 4.3 | SUBJECT EXCLUSION CRITERIA | |
| | | SUBJECT EXCLUSION CRITERIA | 13 |
| | 4.4 | SUBJECT WITHDRAW / EARLY TERMINATION | |
| 5 | | | 13 |
| 5 | | SUBJECT WITHDRAW / EARLY TERMINATION | 13 |
| 5 | STU | SUBJECT WITHDRAW / EARLY TERMINATIONIDY PROCEDURE | 13<br>14<br>14 |
| 5 | STU<br>5.1 | SUBJECT WITHDRAW / EARLY TERMINATION IDY PROCEDURE ENROLLMENT | 13<br>14<br>14 |
| 5 | STU<br>5.1<br>5.1. | SUBJECT WITHDRAW / EARLY TERMINATION | 13<br>14<br>14<br>14 |
| 5 | 5.1<br>5.1.<br>5.2 | SUBJECT WITHDRAW / EARLY TERMINATION IDY PROCEDURE ENROLLMENT 1 INFORMED CONSENT DEMOGRAPHIC AND BASELINE DATA | 13<br>14<br>14<br>14<br>14 |
| 5 | 5.1<br>5.1.<br>5.2<br>5.3 | SUBJECT WITHDRAW / EARLY TERMINATION | 1314141415 |
| 6 | 5.1<br>5.1.<br>5.2<br>5.3<br>5.4<br>5.5 | SUBJECT WITHDRAW / EARLY TERMINATION | 131414141515 |
| | 5.1<br>5.1.<br>5.2<br>5.3<br>5.4<br>5.5 | SUBJECT WITHDRAW / EARLY TERMINATION | 13141414151515 |
| | 5.1<br>5.1.<br>5.2<br>5.3<br>5.4<br>5.5 | SUBJECT WITHDRAW / EARLY TERMINATION | 1314141415151516 |



SPONSOR: ZMS


| 7 | RISK | (S & B | ENEFITS | . 16 |
|---|---|---|---|---|
| | 7.1 | RISK | DETERMINTATION & REDUCTION | . 16 |
| | 7.2 | BEN | EFITS | . 17 |
| 8 | SAFI | ETY A | SSESSMENT AND MANAGEMENT | . 17 |
| | 8.1 | SAFE | TY DEFINITIONS | . 17 |
| | 8.1. | 1 | ADVERSE EVENT (AE) | . 17 |
| | 8.1. | 2 | SERIOUS ADVERSE EVENT (SAE) | . 18 |
| | 8.1. | 3 | UNANTICIPATED ADVERSE DEVICE EFFECT (UADE) | . 18 |
| | 8.2 | SAFE | TY REPORTING | . 19 |
| | 8.2. | 1 | REPORTING EVENTS & SAFETY CONTACTS | . 19 |
| 9 | STA | TISTIC | CAL METHODS AND CONSIDERATIONS | . 19 |
| | 9.1 | SAM | PLE SIZE DETERMINATION | . 19 |
| | 9.2 | DAT | ASETS ANALYZED | . 20 |
| | 9.3 | STAT | FISTICAL ANALYSIS | . 20 |
| | 9.3. | 1 | Descriptive Statistics | . 20 |
| | 9.3. | 2 | STATISTICAL METHOD FOR CONTINUOUS VARIABLES | . 20 |
| | 9.3. | 3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | . 20 |
| | 9.3. | 4 | PRIMARY ANALYSIS | . 20 |
| 10 | <b>)</b> D | ATA ( | COLLECTION, RETENTION, AND MONITORING | .21 |
| | 10.1 | DAT | A COLLECTION | .21 |
| | 10.1 | 1 | SUBJECT CONFIDENTIALITY | .21 |
| | 10.2 | DAT | A RETENTION | . 22 |
| | 10.3 | MON | NITORING | . 22 |
| | 10.3 | 3.1 | MONITORING PLAN | . 22 |
| 1: | L S | TUDY | ADMINISTRATION | .22 |
| | 11.1 | AUD | ITS AND INSPECTIONS | . 22 |
| | 11.2 | PRO | TOCOL AND ICF AMENDMENTS | . 22 |
| | 11.3 | PRO | TOCOL DEVIATIONS | . 22 |
| 12 | 2 E | THICA | AL AND OTHER REGULATORY CONSIDERATIONS | .23 |
| | 12.1 | INST | TTUTIONAL REVIEW BOARD (IRB) REVIEW | . 23 |
| | 12.2 | WRI | TTEN INFORMED CONSENT | .23 |



| SPONSOR: | ZMS |
|----------|-----|
|----------|-----|


| 13 | REFERENCES | 24 |
|----|----------------------------------------|----|
| 14 | ABBREVIATIONS AND DEFINITIONS OF TERMS | 25 |



SPONSOR: ZMS


#### **FIGURES AND TABLES**

| Figure 1: Procedure Overview | 14 |
|--------------------------------------------------------------------|----|
| Table 1: Adverse Event Severity Grading | 17 |
| Table 2: Adverse Events Action(s) Taken | |
| Table 3: Adverse Event Relationship to Donation or Study Procedure | 18 |
| Table 4: Adverse Event Outcome | 18 |
| Table 5: Study Reporting Contacts | 19 |
| Table 6: Abbreviations and Definition of Terms | 25 |



SPONSOR: ZMS


#### **1** INTRODUCTION

Intraoperative and postoperative hemorrhage incidence can vary depending on the type of surgery and can lead to severe clinical complications ranging from mild anemia to fatal hemorrhagic shock. Those that recover from severe hemorrhagic events often have poor functional outcomes and are at risk for greater long-term mortality. Numerous studies reveal that post-operative hemorrhagic events are also quite frequent, occurring in as many as 13 to 19% of patients following various type of surgeries (i.e., major pancreatic resections, transoral robotic surgery (TORS) for oropharyngeal squamous cell carcinoma, and living-donor transplants). Hemorrhagic shock is also a leading cause of death in trauma.<sup>1-6</sup>

Monitoring and detecting fluid changes in patients can be complicated. Physiological responses associated with hemorrhagic events are often delayed because of compensation mechanisms that act to sustain blood pressure and protect tissue perfusion. The ability to continuously and non-invasively detect changes in central blood volume and blood loss will permit appropriate hemodynamic management during events at high risk for acute blood loss such as surgery, trauma, post-operative care and other therapeutic procedures. Through early detection and improved hemodynamic monitoring, optimization of fluid balance, anesthesia titration, and augmenting other acute care management requirements, a clinician should be able to improve overall patient stability, minimize complications, diminish surgical trauma and reduce recovery time.

Current methods for acutely monitoring blood volume and blood loss include monitoring of vital signs (such as heart rate, blood pressure, respirations, and oxygen saturation), invasive central venous (right heart central venous pressure measurement and Swan-Ganz pulmonary capillary wedge pressure measurements) and arterial catheters designed to monitor hemodynamic status centrally. Vital sign monitoring may not indicate small amounts of acute blood loss and arterial and venous cannulations can create insertion complications such as perforations in the vasculature, pneumothorax, arrhythmias, thrombosis and infection. While invasive central monitoring may provide extremely accurate information, changes may not be good indicators of early central hypovolemia or with smaller blood volume reductions<sup>1-2</sup>. New non-invasive technologies have recently become available but often include many physiological parameters that may require expedited clinical interpretation in high stress environments and have not become well-established.

The Zynex Fluid Monitoring System, Model CM-1600 uses a relative patient standard approach by non-invasively and simultaneously monitoring five (5) physiological parameters, including bioelectrical impedance, ECG amplitude, photoplethysmogram (PPG) amplitude, heart rate, and skin temperature. The CM Device starts by creating a baseline for each patient in a normal state. When the monitoring session starts, each patient starts with a Relative Index of 100, signifying the collection of parameters near their original baseline value(s). The Relative Index value acts as a combinational score for all the parameters indicative of relative fluid change. There are two (2) models of the CM Device, Model 1500 (CM-1500) and 1600 (CM-1600) which measure the same five (5) parameters and utilize the same algorithm to output the Relative Index value.




SPONSOR: ZMS


#### 1.1 CLINICAL RATIONALE

The proposed clinical study is designed to validate that the Zynex non-invasive monitoring system (CM-1600) can track blood volume changes in healthy individuals consented to undergo a blood donation. An initial feasibility study was conducted (n = 12 subjects) to confirm that the CM-1500 can be used to track acute blood loss in healthy individuals donating 500mL of blood. Additional studies are being conducted in various healthy volunteer and clinical settings to characterize RI performance when known volumes of fluid are removed. A larger study is necessary with comparative physiological variables to validate the specificity and sensitivity of the CM-1600 in detecting blood loss.

#### 2 INVESTIGATIONAL PLAN

#### 2.1 OBJECTIVES

The primary objective of the study is to determine the specificity and sensitivity of the CM-1600 in detecting minor blood loss as compared to standard physiological parameters.

Exploratory objectives of the study will include:

- Characterize the differences in the relative changes in right vs left antecubital blood donations
- Investigate any possible correlations between adverse events, subject demographics, changes in the Relative Index, and timing of when the events occurred

#### 2.2 STUDY DURATION

Enrollment in the study is expected to take approximately six (6) months, and data analysis may take up to an additional two (2) months to complete.

#### 2.3 STUDY DESIGN

The study is a prospective, non-randomized, non-blinded, non-significant risk, multi-center study enrolling up to 500 healthy adult subjects consented to undergo a whole blood donation procedure.

The present study will involve enrolling subjects that will undergo blood donation wearing the study device (CM-1600) and capture study-required physiological parameters pre-, during, and post-donation.

#### 2.4 STUDY ENDPOINTS

The study endpoints include the change and percentage of change between measurements before and after blood donation in the Relative Index and standard physiological parameters. The change is defined as the value after donation minus the one before donation. The percentage of change is the change value divided by the value before donation. Other endpoints such as area under receiver operating characteristic (ROC) together with sensitivity and specificity at various thresholds are also derived for the Relative Index and each of standard physiological parameters in detecting in detecting minor blood loss (i.e., 450 ml).



SPONSOR: ZMS


#### **3** STUDY DEVICES

#### 3.1 FLUID MONITORING SYSTEM, MODEL CM-1600

#### 3.1.1 DEVICE DESCRIPTION

The CM-1600 is a non-invasive monitoring device predicated by the CM-1500 that simultaneously monitors five (5) parameters of a patient's body. Parameters include bioelectrical impedance, heart rate, ECG amplitude, PPG amplitude, and skin temperature. A combination of these parameters is represented by a single number known as the Relative Index value. This value is indicative of relative changes in fluid volume. The Relative Index is a unique functionality of the Zynex Fluid Monitoring System.

#### 3.1.2 DEVICE DESIGN AND COMPONENTS

The CM-1600 is an all-inclusive device that includes the following components: display monitor (1), power supply (1), wrist wearable (1), wrist strap (1), and electrode array set (2). The electrode array sets are single-use, single-subject.

#### 3.1.3 PRINCIPLES OF OPERATION

The CM-1600 measures bioelectrical impedance (ohms), heart rate (BPM), ECG amplitude, PPG amplitude, and skin temperature (°C or °F). As parameters change, towards indications of fluid change/imbalance, the Relative Index, which acts as a combinational score of percent change values for all of the parameters, will compound these changes into a singular value to signify overall fluid changes/imbalances within the patient's body. When the monitoring session starts, every patient will start with a Relative Index of 100, signifying the combination of physiological parameters is near or at their original baseline values for all five (5) monitored parameters. All parameters are continuously measured and tracked during a monitoring session.

#### 3.1.4 INDICATIONS FOR USE

Per the device's FDA 510(k) submission, the CM-1600 is indicated for monitoring bioelectrical impedance, heart rate, ECG amplitude, and PPG amplitude and their relative changes, indicative of relative changes in fluid volume in adult patients.

#### 3.1.5 INTENDED USE

Per the device's FDA 510(k) submission, the CM-1600 is intended to be used in professional medical environments, i.e., hospitals, clinics, and research institutions. The CM-1600 is a standalone device intended for desktop use, where device operation is to be performed as uninterrupted patient monitoring. The CM-1600 shall only be used by a qualified and trained device operator. The device does not report any diagnosis but provides numerical values; it is ultimately the Investigator's responsibility to make proper diagnosis and judgments based on these values.



SPONSOR: ZMS


#### 4 SUBJECT POPULATION AND SELECTION

#### 4.1 POPULATION AND ANTICIPATED NUMBER OF SUBJECTS

Up to 500 healthy adult subjects who meet the inclusion and exclusion criteria will be enrolled in the study to ensure data from 455 treatment subjects are available for analysis.

#### 4.2 SUBJECT INCLUSION CRITERIA

- I.1 Ability to provide written informed consent
- 1.2 Ability and willingness to comply with the study procedures and duration requirements
- I.3 18 years of age or older
- 1.4 Consented and eligible to undergo a single unit whole blood donation

#### 4.3 SUBJECT EXCLUSION CRITERIA

- E.1 Females who are pregnant or breastfeeding
- E.2 Undergone an amputation of any upper extremity
- E.3 Diagnosed with dextrocardia
- E.4 Subjects who have a pacemaker
- E.5 Subjects with body hair density which prevents adequate application of device electrodes

#### 4.4 SUBJECT WITHDRAW / EARLY TERMINATION

Subjects who withdraw from the study before using the CM-1600 device will be replaced. The reason the subject withdrew from the study may be recorded; subjects are not required to provide a reason. Subject withdrawal / early termination criteria may include but are not limited to:

- W.1 Subject requests to be withdrawn from the study or withdraws consent.
- W.2 Subject refuses to comply with required study procedures.
- W.3 An Adverse Event ("AE") makes the continuation of the subject impossible or inadvisable
- W.4 The Investigator determines it is in the subject's best interest to discontinue from the study.



SPONSOR: ZMS


#### 5 STUDY PROCEDURE

Figure 1: Procedure Overview



#### 5.1 ENROLLMENT

A subject will be considered enrolled in the study after provided written informed consent. Subjects will only be eligible to participate in the study if they have consented to donate one unit of whole blood per the standard of care donation procedures. Enrollment in the study will increase a subject's blood donation duration by approximately 15 minutes.

#### 5.1.1 INFORMED CONSENT

The Investigator or qualified designated study personnel will complete the Informed Consent process before any study procedures may occur. The subject will be provided an IRB-approved version of the Informed Consent Form (ICF). The subject will have an ample amount of time to read the ICF and ask questions before providing written consent. The subject will receive a signed copy of the ICF. The Investigator or qualified designated study personnel will record that consent was obtained prior to performing study procedures.

#### 5.2 DEMOGRAPHIC AND BASELINE DATA

Demographic and enrollment data collection will include obtaining health screening data directly from the standard blood donation screening record at the study site. Data not available on the blood donation procedure record will be captured on a case report form (CRF). These data will include but are not limited to skin tone, smoking history, a blood donation anxiety questionnaire, blood donation history, and if subjects are currently taking any medications or supplements that could impact their physiological response to the donation procedure. Female subjects will self-report they are not currently pregnant or have been pregnant in the previous six (6) weeks, and that will be captured on the standard blood donation screening record.




SPONSOR: ZMS


Baseline hemoglobin will be collected as part of the standard blood donation procedure via a finger stick (or per standard of care for the site). Subjects that are unable to proceed with the blood donation due to their baseline hemoglobin level will be withdrawn from the study.

Following demographic and enrollment data collection and PRIOR to blood donation, all subjects will be connected to the CM-1600 per the Instructions for Use. Designated study personnel must ensure that the subject ID number and gender is entered for each subject prior to starting a new monitoring session.

The CM-1600 will be connected to the subject's left side of the body. The device will be turned on with the subject placed in a resting supine position for a minimum of five (5) minutes before the baseline measurements will be recorded. After the five (5) minute waiting period, study personnel will record, at a minimum, the following: blood pressure, heart rate, respiratory rate, and Relative Index from the CM-1600.

#### 5.3 SUBJECT PARTICIPATION

Subjects will proceed with their blood donation procedure wearing the CM-1600. Immediately prior to the start of the blood donation procedure, the Investigator or designated study personnel will press the "MARK EVENT" button on the CM-1600 which will signify the start of the procedure on the device.

The Investigator or designated study personnel will monitor the subject per standard of care throughout the donation procedure and record any adverse events noted. Total amount of blood collected will vary per subject based upon their estimated blood volume, and the final amount donated will be recorded.

Immediately following completion of the blood donation, the Investigator or designated study personnel should press "EVENT" on the CM-1600. The same physiological parameters collected at baseline will be repeated.

Subjects will remain connected to the CM-1600 for at least ten (10) minutes following the donation procedure. Following the 10-minute post-donation monitoring period, the physiological parameters will be captured one final time, subjects will be disconnected from the study device, and study participation will be complete.

#### 5.4 ADVERSE EVENTS

Adverse Events (AE), Serious Adverse Events (SAE), or Unanticipated Adverse Device Effect (UADE) that occur after informed consent and before completion of the study will be recorded. SAE's may require follow-up contact via a telephone call, depending on the nature of the SAE.

#### 5.5 SUBJECT COMPLETION

Subjects' participation in the study will be considered complete once the monitoring session has ended and the device has been removed.



SPONSOR: ZMS


#### **6** DEVICE MANAGEMENT

#### 6.1 UNPACKING AND INSPECTION

It is the responsibility of the Principal Investigator (PI) to ensure that all study devices are unpacked and inspected prior to using in any study procedures. Upon arrival, the Investigator or designated study personnel will remove the device display monitor and accessories from the shipping container; ensure all device components are received. The study site must inform the Sponsor of any missing or damaged items within seven (7) days. Devices with any missing or damaged items cannot be used and shall be replaced.

#### 6.2 ACCOUNTABILITY, STORAGE & DISPENSATION

It is the responsibility of the Principal Investigator to ensure all study devices are inventoried and accounted for throughout the conduct of the study. The Investigator or qualified designated study personnel will record all information on the Device Accountability forms maintained in the Investigator Site Files (ISF).

The investigational device will be stored at the study center. When not in use, the device will be stored in a secure location (i.e., area with limited access or in a locked cabinet) under appropriate environmental conditions found in the Instructions for Use (IFU) manual.

The study device shall only be used under the supervision of the Principal Investigator or designated study personnel on authorized study subjects.

#### 6.3 CLEANING & RETURN

The study devices shall be cleaned before each use. Cleaning procedures will be followed per the Instructions for Use (IFU) manuals. The study devices and any unused accessories will be returned to the Sponsor after study completion.

#### 7 RISKS & BENEFITS

#### 7.1 RISK DETERMINTATION & REDUCTION

This study is determined to be non-significant risk. An Investigational Device Exemption will not be submitted based on this determination.

Study subjects are subject to risk no greater than or similar to risks associated with undergoing a blood donation. The use of the CM-1600 does not meet the definition of significant risk under 21CRF 812.3 (m). All adverse events will be recorded and analyzed to evaluate their significance. Possible risks may include:

- [Possible, Rare] Skin irritation could occur from the electrodes
- [Possible, Mild] Discomfort could occur due to lying in a supine position for duration of the donation procedure.




SPONSOR: ZMS


Every possible effort will be made to reduce the risks to a minimum. Investigators or qualified designated study personnel will be experienced and skilled in blood donation procedures, receive training on the protocol and use of the device. All adverse events will be documented and reported to the Sponsor.

#### 7.2 BENEFITS

This study is for research purposes only. There is no direct benefit to subjects participating in the study. Information from this study may help other people in the future.

#### **8** SAFFTY ASSESSMENT AND MANAGEMENT

Safety will be assessed by reviewing and summarizing adverse events.

#### 8.1 SAFETY DEFINITIONS

#### 8.1.1 ADVERSE EVENT (AE)

An Adverse Event (AE) is defined as any untoward medical occurrence, whether or not related to the study device or study procedure. AE's are characterized by grading, actions taken, relationship to donation or study procedure, and outcome. These definitions are in the corresponding tables below. All adverse events related to the blood donation procedure will be recorded and reported in addition to those that may occur specific to the protocol-defined study procedure. All attempts should be made to ensure resolution of the adverse event upon study completion.

Table 1: Adverse Event Severity Grading

| Severity | Description |
|---|---|
| Grade 1: Mild | Awareness of signs or symptoms, but they are easily tolerated |
| Grade 2: Moderate | Enough discomfort to cause interference with usual activity |
| Grade 3: Severe | Incapacitating, with the inability to work or do usual activity |
| Grade 4: Fatal | Subject expired/death occurred |

Table 2: Adverse Events Action(s) Taken

| Action Taken<br>(Check all that apply) | Description |
|---|---|
| None | No actions were taken, observation only. |
| Medications | Subject required medication(s) |
| Other Treatment | Subject required other treatment(s) |
| Early Withdrawal | Adverse event led to early study withdrawal |



SPONSOR: ZMS


Table 3: Adverse Event Relationship to Donation or Study Procedure

| Relationship | Description |
|---|---|
| None | Causal relationship can be ruled out |
| Possible – Donation Procedure | Causal relationship is reasonably possible to the blood donation |
| | procedure (i.e., the relationship cannot be ruled out) |
| Bassible Church Basics | Causal relationship is reasonably possible to the study device (i.e., |
| Possible – Study Device | the relationship cannot be ruled out) |
| Yes – Donation Procedure | Causal relationship to the donation procedure is certain |
| Yes – Study Device | Causal relationship to the study device is certain |

Table 4: Adverse Event Outcome

| Outcome | Description |
|---|---|
| Recovered/Resolved | Subject recovered and event was resolved upon study completion |
| Recovered/Resolved with | Subject recovered but exhibited lingering minor symptoms upon |
| Sequelae | study completion |
| Recovering | Adverse event persisted upon study completion but was improving |
| Not Decemend | Adverse event persisted upon study completion and was not |
| Not Recovered | exhibiting any signs of improvement |
| Death | Subject expired |
| Unknown | Status of the adverse event was unknown upon study completion |

#### 8.1.2 SERIOUS ADVERSE EVENT (SAE)

An SAE is defined as an AE that meets any of the following criteria: Fatal or life-threatening\*; requires or prolongs in-subject hospitalization\*\*; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical event. An event's severity grading, action(s) taken, relationship to the donation or study procedure, and the outcome will all be used for SAE's.

#### 8.1.3 UNANTICIPATED ADVERSE DEVICE EFFECT (UADE)

An unanticipated adverse device effect is defined by 21 CFR 812.3 as any serious adverse effect on the health of safety or life-threatening problem or death caused by or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including supplementary plan or application, or any other unanticipated serious problem associated with the device that relates to the rights, safety, or welfare of

<sup>\*</sup>Life-threatening is defined as an event in which the subject was at risk of death at the time of the event. It does not refer to an event that hypothetically may have caused death if it was more severe.

<sup>\*\*</sup>In-subject hospitalization is defined as an event in which the subject was admitted to the hospital for one or more days, even if released on the same day or an emergency room visit, which results in admission to the hospital. Emergency room visits that do not result in admission to the hospital should be evaluated for one of the other serious outcomes criteria.



SPONSOR: ZMS


subjects. The Investigator or designee will indicate if they believe an event was an unanticipated adverse device effect on the case report form, and the Sponsor will evaluate for reporting requirements defined below.

#### 8.2 SAFETY REPORTING

Safety reporting begins at the time of signed Informed Consent and ends at subject study completion.

Investigators shall submit to the Sponsor a report of any AE's or SAE's that occur during the study within five (5) working days but no later than ten (10) days after the Investigator learns of the event.

Investigators shall submit to the Sponsor a report of any UADE(s) that occur during the study as soon as possible but no later than five (5) working days after the Investigator learns of the effect. Sponsors will evaluate UADE's.

#### 8.2.1 REPORTING EVENTS & SAFETY CONTACTS

Events will be reported, in writing, to the Sponsor as soon as possible but no later than five (5) working days after the Investigator learns of the event. In an event resulting in the death of the subject, the event will be reported within 24-hours of knowledge of the event. The Sponsor is responsible for fulfilling IRB and regulatory reporting requirements.

Contact Contact Information

Zynex Monitoring Solutions

WCG IRB

WCG IRB

Zynex Monitoring Solutions

Attn: ZMS Clinical
9555 Maroon Circle
Englewood, CO 80112

**Table 5: Study Reporting Contacts** 

#### 9 STATISTICAL METHODS AND CONSIDERATIONS

#### 9.1 SAMPLE SIZE DETERMINATION

This study is designed to evaluate the sensitivity and specificity of the CM Device in detecting minor blood loss as compared to standard physiological parameters. The sample size was calculated based on the following assumptions:

1) Standard deviation for the decrease after blood donation using the CM-1600 = 6.5 RI units




SPONSOR: ZMS


- 2) Minimum detectable difference after the donation = 1 RI unit
- 3) Power 90% and one-sided alpha = 0.025

A sample size of 455 will achieve about 90% power to detect a minimum difference of interest 1.0 RI unit with an estimated standard deviation of 6.5 and with a significance level (alpha) of 0.025 using a one-sided one-sample t-test.

To adjust for possible attrition or incomplete datasets/donations, 10% has been added to the sample size, therefore, a total of 500 subjects will be enrolled.

#### 9.2 DATASETS ANALYZED

All eligible subjects who were enrolled in the study and connected to the study devices will be included in the analyses. Subjects who withdraw after enrollment and before the study devices are connected will be excluded from the analyses.

#### 9.3 STATISTICAL ANALYSIS

#### 9.3.1 Descriptive Statistics

Continuous data will be summarized in terms of the mean, standard deviation (SD), median, quartiles, minimum, maximum, and number of observations, unless otherwise specified. Categorical data will be summarized in terms of the number of subjects providing data at the relevant time point (n), frequency count, and percentage. Percentages will be calculated using n as the denominator.

#### 9.3.2 STATISTICAL METHOD FOR CONTINUOUS VARIABLES

The normality of continuous data will be assessed both visually and by Shapiro-Wilk test. If data are considered normally distributed, the 95% CI of the mean will be constructed based on a t-distribution. Otherwise, if data are skewed, distribution-free confidence interval of the median will be calculated. The comparison between before and after blood donation will be conducted by using paired t-test or Wilcoxon signed-rank test, depending on the distribution of data.

#### 9.3.3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

All baseline demographic variables collected at enrollment will be summarized using descriptive statistics.

#### 9.3.4 PRIMARY ANALYSIS

The following will cover the planned primary analyses for this study procedure. Unless otherwise specified, statistical analyses will be performed using two-sided hypothesis tests at the overall 5% significance level. No multiple comparison adjustments will be performed.

1. Analysis of measurements taken before and after blood donation

Measurements including RI and individual physiological parameters taken before and after blood donation will be first summarized using descriptive statistics. For each parameter, the absolute and percent differences before and after donation will be calculated and summarized using summary statistics



SPONSOR: ZMS


together with 95% confidence interval. The p-value will be calculated using paired t-test or Wilcoxon signed-rank test to compare with zero.

2. Analysis of differences between measurement taken before and after blood donation.

The difference between measurement taken before and after blood donation will be calculated by value before donation minus value after donation for RI and each individual physiological parameter.

#### 3. ROC Analysis

Receiver operator characteristic (ROC) will be used to evaluate the sensitivity and specificity at various cutoff points in detecting one Unit (approximate 450mL) blood loss (donation) using the RI. The ROC curves will be plotted using the data collected before and after donation, and the areas under the curves (AUCs) will be derived together with a 95% confidence interval using an asymptotic approach. The ROC curves will be constructed for the percentage of decreases between RI measured before and after blood donation against the one Unit blood donation. Similar ROC analyses will be also conducted for each of the individual physiological parameters. These ROC curves will be plotted in an overlay format to demonstrate the difference in the detection of blood loss in the various parameters and indices.

Several cutoff points will be chosen to compare sensitivity, specificity, positive predictive value, negative predictive value, and positive and negative likelihood ratios.

# 10 DATA COLLECTION, RETENTION, AND MONITORING

#### 10.1 DATA COLLECTION

The Investigator will prepare, maintain, and retain complete, current, accurate, organized, and legible Source Documents to record all observations and other pertinent data for each subject. In some instances, case report forms (CRFs) will serve as source documentation. The Investigator or designated study personnel will provide the Sponsor redacted standard procedure records with the subject ID number as applicable. Any required data not collected as standard of care for the blood draw procedure will be captured on study-specific case report forms.

Corrections of data on paper source documents will be made by crossing out the incorrect data and making the GCP-compliant correction. Each correction will be initialed and dated by the study personnel making the correction.

The Investigator is responsible for the information collected on subjects enrolled in the study. All data collected during the study must be reviewed and verified for completeness and accuracy by the Investigator. If any corrections are made after the Investigators signature, the Investigator will also initial and date the correction.

#### 10.1.1 SUBJECT CONFIDENTIALITY

In order to maintain subject confidentiality, records identifying the subject will be kept in a safe and secure location; access to these records will be on a limited basis. Only the subject identification number, gender,



SPONSOR: ZMS


and age will identify study subjects on CRFs and other documentation submitted to the Sponsor. A limited number of Sponsor representatives may have access to identifiable information and will take reasonable precautions to maintain the confidentiality of the subject's identity.

#### 10.2 DATA RETENTION

All study records will be stored in a safe and secure location. Records will be retained per applicable regulatory requirements, which include for a period of two (2) years after the latter of the following two days: the date which the investigation is terminated or completed, or the date that records are no longer required for purposes of supporting premarket approval applications or a notice of completion of a product development protocol. The Investigator site may transfer custody or records to the Sponsor with appropriate documentation recording the transfer.

#### 10.3 MONITORING

#### 10.3.1 MONITORING PLAN

Monitoring visits will be conducted by representatives of the Sponsor or study site or both according to 21 CFR 812. (c) for non-significant risk device studies and ICH Guidelines. By signing this protocol, the Investigator grants permission to the Sponsor (or designee) and all appropriate regulatory authorities to conduct on-site or electronic monitoring or auditing or both of all appropriate study documentation.

#### 11 STUDY ADMINISTRATION

#### 11.1 AUDITS AND INSPECTIONS

External auditors and government inspectors may evaluate the study and must be allowed access to CRFs, source documents, and other study files. Audit reports will be confidential.

#### 11.2 PROTOCOL AND ICF AMENDMENTS

Sponsor approval is required for any protocol or ICF amendment. Protocol or ICF amendments will not be implemented without prior written IRB approval except as allowed per the IRB procedures/approval and as necessary to eliminate immediate safety hazards to subjects. A protocol amendment intended to eliminate an apparent immediate hazard to subjects may be implemented immediately, provided IRBs are notified within five (5) working days. The Informed Consent Form will be reviewed and updated as necessary at the time of the protocol amendment.

#### 11.3 PROTOCOL DEVIATIONS

A protocol deviation is defined as any accidental or unintentional changes to, or non-compliance with the IRB approved research protocol. Any deviation from the protocol must be documented and reported to the Sponsor within ten (10) working days and reported to the IRB as applicable to regulatory requirements. Protocol deviations that pose an immediate risk or significant hazard to subjects must be reported to the Sponsor within 24 hours and reported to the IRB no later than five (5) working days after the emergency occurred. In the instance an Investigator uses a device without obtaining informed



SPONSOR: ZMS


consent; the Investigator shall report to the Sponsor and the IRB within five (5) working days as per 21 CFR 812.150 (1) (5).

### 12 ETHICAL AND OTHER REGULATORY CONSIDERATIONS

It is the responsibility of the Investigator that the study is conducted according to the Declaration of Helsinki, Protection of Human Volunteers (21 CFR 50), Institutional Review Board (21 CFR 56), and Responsibilities of Clinical Investigators (21 CFR 812 (e)).

#### 12.1 INSTITUTIONAL REVIEW BOARD (IRB) REVIEW

The Protocol, ICF, and any subject facing material (as required) will be reviewed and approved by the IRB prior to study initiation. The Sponsor will maintain responsibility for obtaining IRB approval and submitting all required study reports to the IRB. Amendments to the Protocol, ICF, or any subject facing material will not be implemented without prior written IRB approval unless to eliminate an apparent immediate hazard to subjects. All IRB approvals will be kept in the Trial Master File and Investigator Site File.

#### 12.2 WRITTEN INFORMED CONSENT

The Informed Consent Form (ICF) and Informed Consent process will include all elements required by applicable regulations. Informed consent will be obtained in accordance with the Declaration of Helsinki, ICH, Good Clinical Practice, and US Code of Federal Regulations for Protection of Human Subjects (21 CFR 50.25 [a,b], 21 CFR 50.27, and 21 CFR Part 56, Subpart A), the Health Insurance Portability and Accountability Act (HIPAA) when applicable, and local regulations.

A properly executed, written informed consent will be obtained from all subjects prior to entering the subject into the trial, unless waived by the IRB. ICF information will be given in both verbal and written form. The subject must be given an ample amount of time to read the ICF. The subject must provide written consent by signing and dating the approved ICF. A signed copy of the ICF will be provided to the subject; originals will be maintained with the subject's study records.

Assents Forms will not be permitted as subjects must be over the age of 18 to meet the Inclusion/Exclusion criteria. Legally Authorized Representatives will not be permitted as subjects must have the ability to provide written consent to meet the Inclusion/Exclusion criteria.

# ZYNEX

# **CLINICAL PROTOCOL**

SPONSOR: ZMS


#### 13 REFERENCES

1 Little R, Kirkman E, Driscoll P, Hanson J, Mackay-Jones K. Preventable Deaths after Injury: Why are the Traditional "Vital" Signs Poor Indicators of Blood Loss. Journal of Accident and Emergency Medicine. 1995;12: 1-14.

2 Convertino VA, Moulton SL, Grudic GZ, Rickards CA, Hinojosa-Laborde C, Gerhardt RT, et al. Use of advanced machine-learning techniques for noninvasive monitoring of hemorrhage. The Journal of trauma. 2011;71(1 Suppl):S25-32.

3 Ansari D, Tingstedt B, Lindell G, Keussen I, Ansari D, Andersson R. Hemorrhage after Major Pancreatic Resection: Incidence, Risk Factors, Management, and Outcome. Scand J Surg. 2017;106(1):47-53. doi:10.1177/1457496916631854

4 Kubik M, Mandal R, Albergotti W, Duvvuri U, Ferris RL, Kim S. Effect of transcervical arterial ligation on the severity of postoperative hemorrhage after transoral robotic surgery. Head Neck. 2017;39(8):1510-1515. doi:10.1002/hed.24677

5 Hsieh CE, Chou CT, Lin CC, et al. Hemodynamic Changes Are Predictive of Coagulopathic Hemorrhage After Living Donor Liver Transplant. Exp Clin Transplant. 2017;15(6):664-668. doi:10.6002/ect.2016.020

6 Frank SM, Savage WJ, Rothschild JA, Rivers RJ, Ness PM, Paul SL, et al. Variability in blood and blood component utilization as assessed by an anesthesia information management system. Anesthesiology. 2012;117(1):99-106.



SPONSOR: ZMS


# **14** ABBREVIATIONS AND DEFINITIONS OF TERMS

Table 6: Abbreviations and Definition of Terms

| Abbreviation | Definition |
|-----------------|---------------------------------------------------------|
| AE | Adverse event |
| BPM | Beats per minute |
| BP | Blood pressure |
| С | Celsius |
| CFR | U.S. Code of Federal Regulations |
| CM-1500/CM-1600 | Zynex Fluid Monitoring System, Model 1500 or Model 1600 |
| CRF | Case report form |
| ECG | Electrocardiogram |
| e.g. | Exempli Gratia (for example) |
| F | Fahrenheit |
| FDA | U.S. Food and Drug Administration |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | Heart rate |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonization |
| IFU | Instructions for Use |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| ISO | International Organization for Standardization |
| lb | Pound; unit of mass |
| ohms | Plural unit of electrical resistance |
| mL | Milliliter |
| PHI | Protected Health Information |
| PI | Principal Investigator |
| PPG | Photoplethysmogram |
| SAE | Serious adverse event |
| UADE | Unanticipated Adverse Device Event |
| ZMS | Zynex Monitoring Solutions |